CLINICAL TRIAL: NCT00365625
Title: Patient Orientated Basic Science Investigation: Determination of Lymphocyte JAM-C Expression in Patients With Psoriasis Vulgaris
Brief Title: Determination of Lymphocyte JAM-C Expression in Patients With Psoriasis Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Prof. Ralf Ludwig, Johann Wolfgang Goethe University Hospitals
Other Study IDs: 244/06
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-08

CONDITIONS: Psoriasis; Psoriasis Vulgaris
Keywords: Psoriasis; JAM3 protein, human; Cell Adhesion Molecules; Skin; Inflammation; Lymphocytes
MeSH Terms: conditions — Psoriasis; Inflammation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The stepwise process of leukocyte extravasation to inflamed tissues depends on the expression of a variety of cytokines and adhesion molecules. Recently much attention has focused on the Junctional Adhesion Molecules (JAM). The three members of this adhesion molecule family, namely, JAM-A, -B and -C, have been shown to govern the last step of leukocyte extravasation (transmigration) - the process of leukocytes passing between endothelial cells. In addition to transmigration, some members of this family seem to support additional steps in the leukocyte extravasation cascade. The investigators recently showed, that antibody-mediated inhibition of JAM-C significantly reduced hapten induced skin inflammation (J Invest Dermatol;125(5):969).

Recent unpublished work from our laboratory showed, that JAM-C expression of lymphocytes can be up-regulated through specific activators. Hence, the investigators hypothesize, that JAM-C expression is elevated in patients with psoriasis. As it is currently not know, which factors may influence the expression of JAM-C, the investigators intend to analyse JAM-C expression on CD3+CD41- cells at several time-points during the treatment of psoriatic patients. Expression of JAM-C will then be correlated to disease activity (PASI).

DETAILED DESCRIPTION:
The stepwise process of leukocyte extravasation to inflamed tissues depends on the expression of a variety of cytokines and adhesion molecules. Recently much attention has focused on the Junctional Adhesion Molecules (JAM). The three members of this adhesion molecule family, namely, JAM-A, -B and -C, have been shown to govern the last step of leukocyte extravasation (transmigration) - the process of leukocytes passing between endothelial cells. In addition to transmigration, some members of this family seem to support additional steps in the leukocyte extravasation cascade. We recently showed, that antibody-mediated inhibition of JAM-C significantly reduced hapten induced skin inflammation (J Invest Dermatol;125(5):969).

Recent unpublished work from our laboratory showed, that JAM-C expression of lymphocytes can be up-regulated through specific activators. Hence, we hypothesize, that JAM-C expression is elevated in patients with psoriasis. As it is currently not know, which factors may influence the expression of JAM-C, we intend to analyse JAM-C expression on CD3+CD41- cells at several time-points during the treatment of psoriatic patients. Expression of JAM-C will then be correlated to disease activity (PASI).

Detailed in- and exclusion criteria are outlined below.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis vulgaris
* PASI >/= 10 at inclusion

Exclusion Criteria:

* Psoriasis arthritis
* Psoriasis pustulosa
* Psoriasis palmoplantaris
* Pregnancy
* current infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: psoriasis patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2005-07; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf J Ludwig, MD, Principal Investigator — Department of Dermatology - Clinic of the Johann Wolfgang Goethe University; Roland Kaufmann, Professor, Study Chair — Department of Dermatology - Clinic of the Johann Wolfgang Goethe University; Wolf-Henning Boehncke, Professor, Study Chair — Department of Dermatology - Clinic of the Johann Wolfgang Goethe University
Locations (1):
- Department of Dermatology - Clinic of the Johann Wolfgang Goethe University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Ludwig RJ, Zollner TM, Santoso S, Hardt K, Gille J, Baatz H, Johann PS, Pfeffer J, Radeke HH, Schon MP, Kaufmann R, Boehncke WH, Podda M. Junctional adhesion molecules (JAM)-B and -C contribute to leukocyte extravasation to the skin and mediate cutaneous inflammation. J Invest Dermatol. 2005 Nov;125(5):969-76. doi: 10.1111/j.0022-202X.2005.23912.x. PMID 16297198
- [Background] Santoso S, Sachs UJ, Kroll H, Linder M, Ruf A, Preissner KT, Chavakis T. The junctional adhesion molecule 3 (JAM-3) on human platelets is a counterreceptor for the leukocyte integrin Mac-1. J Exp Med. 2002 Sep 2;196(5):679-91. doi: 10.1084/jem.20020267. PMID 12208882
- [Background] Chavakis T, Keiper T, Matz-Westphal R, Hersemeyer K, Sachs UJ, Nawroth PP, Preissner KT, Santoso S. The junctional adhesion molecule-C promotes neutrophil transendothelial migration in vitro and in vivo. J Biol Chem. 2004 Dec 31;279(53):55602-8. doi: 10.1074/jbc.M404676200. Epub 2004 Oct 14. PMID 15485832
- [Background] Muller WA. Leukocyte-endothelial-cell interactions in leukocyte transmigration and the inflammatory response. Trends Immunol. 2003 Jun;24(6):327-34. doi: 10.1016/s1471-4906(03)00117-0. PMID 12810109
- [Background] Vonlaufen A, Aurrand-Lions M, Pastor CM, Lamagna C, Hadengue A, Imhof BA, Frossard JL. The role of junctional adhesion molecule C (JAM-C) in acute pancreatitis. J Pathol. 2006 Aug;209(4):540-8. doi: 10.1002/path.2007. PMID 16767690
- [Background] Santoso S, Orlova VV, Song K, Sachs UJ, Andrei-Selmer CL, Chavakis T. The homophilic binding of junctional adhesion molecule-C mediates tumor cell-endothelial cell interactions. J Biol Chem. 2005 Oct 28;280(43):36326-33. doi: 10.1074/jbc.M505059200. Epub 2005 Aug 23. PMID 16118203
- [Background] Lamagna C, Hodivala-Dilke KM, Imhof BA, Aurrand-Lions M. Antibody against junctional adhesion molecule-C inhibits angiogenesis and tumor growth. Cancer Res. 2005 Jul 1;65(13):5703-10. doi: 10.1158/0008-5472.CAN-04-4012. PMID 15994945
- [Background] Aurrand-Lions M, Lamagna C, Dangerfield JP, Wang S, Herrera P, Nourshargh S, Imhof BA. Junctional adhesion molecule-C regulates the early influx of leukocytes into tissues during inflammation. J Immunol. 2005 May 15;174(10):6406-15. doi: 10.4049/jimmunol.174.10.6406. PMID 15879142